CLINICAL TRIAL: NCT02193230
Title: Taking Into Account the Patient/Parent Preference in the Galenic Choice in Atopic Dermatitis. Feasibility and Impact on Treatment Adherence.
Acronym: DACE
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC14_0073
Record Dates: First submitted 2014-07-15; First posted 2014-07-17 (Estimated); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis, Feasibility, Adherence to treatment
MeSH Terms: conditions — Dermatitis, Atopic; Treatment Adherence and Compliance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Atopic dermatitis is a chronic inflammatory skin disease often occurring in childhood.

The treatment consists in making daily local treatment with topical steroid on inflammatory lesions and emollient on the whole body. However, approximately 70% of patients do not adhere to therapy.

Studies have shown that this treatment failure is caused by the complexity of the treatment, the time required for its implementation, the cost of treatment, the dosage of the products, fear of side effects or misunderstanding about the chronicity of these diseases inflammatory conditions of the skin.

This study aims to evaluate the consideration of patient preference in the choice of excipient used for the topical treatment of eczema.

DETAILED DESCRIPTION:
Day 0 :

* Inclusion, collecting non-opposition
* Presentation of the samples: 4 products presented in the same packaging (pump bottle 200 ml) and ranked in order of their fat content:
* Cold Cream: 88%
* Modified Cerat Galen (national formulary): 66%
* Cold Cream Fluid: 32%
* Ointment: 21% The 4 products are all equally effective and suited in the treatment of atopic dermatitis.

The patient choose the cream it will apply from 4 presented. A total of two bottles will be given to the patient. A bottle containing only the emollient applied to dry areas and another bottle in which 30% will be added Diprosone (topical steroid) to be applied on areas of eczema).

* Remitting the questionnaires
* Severity scoring of atopic dermatitis (SCORAD)

Day 30:

* Remitting the questionnaires
* Treatments delivery for 2 months
* SCORAD / PO SCORAD
* Treatment weighing

Day 90:

* SCORAD / PO-SCORAD
* Treatments weighing
* Remitting the final questionnaire

ELIGIBILITY:
Inclusion Criteria:

Patients experiencing treatment failure despite appropriate treatment. Patients minors aged between 3 and 15 years For children age 7 and non-autonomous children in the application of treatment, the parent at the initial consultation should be the one who treats the child.

Information from both parents or parental authority and collection of Non-Opposition The patient must have a computer to do its PO-SCORAD between consultations. Patient who used a topical treatment for atopic dermatitis in the week preceding the study.

Exclusion Criteria:

Patient refusal to participate in the clinical study. Adults and children over 15 years.

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Multicenter prospective nonrandomized uncontrolled open-label study
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2014-10-14 (Actual); Primary Completion 2015-09-30 (Actual); Study Completion 2015-10-31 (Actual)

PRIMARY OUTCOMES:
Assess the feasibility of giving the choice to the patient/parent of different galenic in atopic dermatitis. | 90 days
  Assess the feasibility of giving the choice to the patient/parent of different galenic in atopic dermatitis.
  The primary outcome is evaluated through a questionnaire given to the patient/parent at day 0 day 30 day 90.

SECONDARY OUTCOMES:
Evaluate the impact of this procedure in patient adherence to treatment (trough weighing treatments at day 30 and day 90) | 90 days
Evaluate the impact of this procedure on the evolution of the disease | 90 days
  Evaluate the impact of this procedure on the evolution of the disease (trough SCORAD and PO-SCORAD at day 0, day 30, day 90)
Assess the feasibility point of view of the prescribing physician | 90 days
  - Assess the feasibility point of view of the prescribing physician (through questionnaires at day 0 day 30 day 90)
Measuring the characteristics of a specified product and those of a product chosen by the patient | 90 days
  - Measuring the characteristics of a specified product and those of a product chosen by the patient (through questionnaires at day 0, day 30, day 90)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Stalder, PU-PH, Study Director — Nantes University Hospital; Jean-Marc Chavigny, PH, Principal Investigator — Centre Pasteur Dermatologie
Locations (1):
- CHU de Nantes, Nantes, France

REFERENCES:
- See also: PO SCORAD — http://www.decas.univ-nantes.fr/GET/GET/POSCORAD_files/Po-Scorad_FR.pdf